CLINICAL TRIAL: NCT04987034
Title: Endoscopic Ultrasound-Guided Portosystemic Pressure Gradient Measurements vs. Transjugular Balloon Occlusion Measurement: A Multicenter EU Study
Brief Title: Comparing a Direct Versus an Indirect Approach to Measuring the Portalsytemic Pressure Gradients
Status: Completed | Type: Observational
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Other Study IDs: 16-11
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Liver Cirrhosis
Keywords: Portal Pressure Measurement; Portal Pressure Gradient; Hepatic Vein Pressure Gradient; Liver Diseases; Portal Hypertension; Intractable ascites; End Stage Liver Disease
MeSH Terms: conditions — Liver Cirrhosis; Liver Diseases; Hypertension, Portal; End Stage Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Direct and indirect PPG measurements: Measuring the portalsystemic pressure gradient in patients directly using the EchoTip® Insight™ and indirectly through the HVPG procedure.
  Interventions: Device: EchoTip® Insight™

INTERVENTIONS:
Device: EchoTip® Insight™ — Patients will undergo procedure where HVPG is obtained under mild sedation, next the patients will undergo anesthesia and mechanical intubation where HVPG measurements will be obtained simultaneously with the EchoTip Insight measurement. For patients receiving a transjugular intrahepatic portosystemic shunt (TIPS), direct portal vein pressure measurements will be obtained by the EchoTip® Insight™ and compared to the transjugular direct portal vein measurement obtained during the interventional radiology (IR) procedure.

SUMMARY:
The objective of this study is to evaluate the correlation of the calculated portosystemic pressure gradient (PPG) obtained by direct portal and hepatic pressure measurements with the EchoTip® Insight™ and indirect portal vein pressure measurements using the interventional radiology based hepatic venous pressure gradient (HVPG) procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis who have been referred for a procedure where HVPG is obtained.

Exclusion Criteria:

* Patient is pregnant, breast-feeding, or planning to become pregnant during the course of the study
* Patient is unwilling or unable to sign and date the informed consent
* Patient is unwilling to comply with the follow-up study schedule
* Previous total or partial splenectomy
* Non-cirrhotic portal hypertension
* Known history of spontaneous bacterial peritonitis (SBP) within the last three months irrespective of treatment for SBP
* Patients with known infection which is not controlled by medical intervention
* Portopulmonary hypertension
* Cardiac decompensation
* Pre-sinusoidal liver disease
* Cholestatic liver disease
* Patient who received endoscopic treatment for upper gastrointestinal (GI) variceal bleeding within the past 7 days
* Patients with current hepatocellular carcinoma (HCC)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis who have been referred for a HVPG procedure.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The correlation between the direct and indirect procedures to measure PPG. | The period from the start of the procedure until all measurements are completed is anticipated to be approximately two hours
  Under general anesthesia, to quantify the correlation between the calculated PPG from the EchoTip® Insight™ direct measurements (difference between direct portal vein pressure and direct hepatic vein pressure) and indirect HVPG measurement (difference between transjugular free hepatic venous pressure (FHVP) and wedge hepatic venous pressure (WHVP) obtained during an IR procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Schalk Van der Merwe, Prof, Principal Investigator — Department of Gastroenterology and Hepatology and Department of Clinical and Experimental Medicine
Locations (3):
- University Hospitals Leuven, Leuven, Belgium
- Erasmus University Medical Center, Rotterdam, Netherlands
- Hospital Clinic, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Cook Research Incorporated (CRI) is fully committed to supporting the principles of responsible data sharing, including providing qualified scientific researchers access to deidentified, patient-level data from CRI clinical studies to conduct legitimate scientific research. Data underlying the results reported in this clinical study will be made available for request after final report has been distributed and ending 5 years after final report has been distributed. Interested researchers may review the "Cook Research Incorporated Policy on Access to Clinical Study Data" at https://www.cookresearchinc.com/extranet/data-access.html and submit a complete research proposal to request data access. Additional study documents (such as the study protocol) will be shared as needed if the data access request is granted. A data sharing agreement will be executed for access to deidentified patient-level data.

REFERENCES:
- [Derived] Vanderschueren E, Laleman W, Bonne L, Maleux G, Wagner DR, Yeh C, Calvo A, Sendino O, Gines A, Baiges A, Bruno MJ, Garcia-Pagan JC, van der Merwe S. Endoscopic ultrasound-guided portosystemic pressure gradient measurement vs. transjugular balloon occlusion measurement in patients with cirrhosis (ENCOUNTER): A bicentric EU study. JHEP Rep. 2025 May 29;7(8):101466. doi: 10.1016/j.jhepr.2025.101466. eCollection 2025 Aug. PMID 40689144